CLINICAL TRIAL: NCT06718582
Title: Effect of Limb Occlusion Pressure Attainment on Cardiovascular, Perceptual, and Performance Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Teri Herberger (Other)
Responsible Party: Sponsor-Investigator, Teri Herberger, Director of Sponsored Research Programs, Salisbury University
Organization: Salisbury University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: #430
Record Dates: First submitted 2024-12-02; First posted 2024-12-05 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Blood Flow Restriction (BFR) Training Effects; Arterial Stiffness, Blood Pressure; Muscle Morphology; Perceptions
Keywords: blood flow restriction training; arterial stiffness; rating of perceived effort; traing volume; rating of perceived discomfort

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Supine Limb Occlusion Pressure (Experimental): In the supine LOP session, the BFR cuffs will be pressurized to 60% of the supine LOP. After inflation of the BFR cuffs, four sets of dumbbell wall squats will be performed to failure with a 2-seconds concentric and 2-seconds eccentric cadence, at 20% of their 1RM using 60% of the LOP with 1-minute rest intervals.
  Interventions: Device: Delfi Training Device
- Seated Limb Occlusion Pressure (Experimental): In the seated LOP session, the BFR cuffs will be pressurized to 60% of the seated LOP. After inflation of the BFR cuffs, four sets of dumbbell wall squats will be performed to failure with a 2-seconds concentric and 2-seconds eccentric cadence, at 20% of their 1RM using 60% of the LOP with 1-minute rest intervals.
  Interventions: Device: Delfi Training Device
- Standing Limb Occlusion Pressure (Experimental): In the standing LOP session, the BFR cuffs will be pressurized to 60% of the standing LOP. After inflation of the BFR cuffs, four sets of dumbbell wall squats will be performed to failure with a 2-seconds concentric and 2-seconds eccentric cadence, at 20% of their 1RM using 60% of the LOP with 1-minute rest intervals.
  Interventions: Device: Delfi Training Device
- No BFR cuff (Placebo Comparator): Four sets of dumbbell wall squats will be performed to failure with a 2-seconds concentric and 2-seconds eccentric cadence, at 20% of their 1RM using 60% of the LOP with 1-minute rest intervals with no BFR cuffs
  Interventions: Device: Delfi Training Device

INTERVENTIONS:
Device: Delfi Training Device — Delfi (Vancouver, Canada) training devices will be used for exercise and testing sessions. Cuffs will be placed around the right and left proximal thigh. The LOP will be set at 60% immediately before exercise and will be applied during the entire exercise set (approximately 30-60 seconds in duration) following manufacturer specifications. In the supine LOP session, the BFR cuffs will be pressurized to 60% of the supine LOP. In the seated LOP session, the BFR cuffs will be pressurized to 60% of the seated LOP. And, in the standing LOP session, the BFR cuffs will be pressurized to 60% of the standing LOP. The cuffs will maintain pressure during training and rest periods. The LOP will be reduced to 0% immediately after completing the last set.

SUMMARY:
To test the effect of limb occlusion pressure attainment in the supine, seated, and standing position on exercise performance, vascular physiology, and muscle.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the attainment of limb occlusion pressure (LOP)in the supine, seated, and standing positions on indices of arterial stiffness, muscle morphology, participant perception, and performance responses. Thirty adults aged 18-40 will undergo four treatment sessions (control (no BFR), supine LOP, seated LOP, and standing LOP) in a randomized order separated by one week. A familiarization session will also occur one week before starting the treatment period. Each subject will undergo a series of tests including anthropometry, ultrasonography of the carotid artery, applanation tonometry, ultrasonography of the vastus lateralis, blood pressure acquisition, body composition, and maximal strength assessments (1RM). All sessions will consist of four sets of dumbbell wall squats performed to failure with a 2-seconds concentric and 2-seconds eccentric cadence, at 20% of their 1RM using 60% of the LOP with 1-minute rest intervals. In the supine LOP session, the BFR cuffs will be pressurized to 60% of the supine LOP. In the seated LOP session, the BFR cuffs will be pressurized to 60% of the seated LOP. And, in the standing LOP session, the BFR cuffs will be pressurized to 60% of the standing LOP. Assessments will be performed immediately before and after the exercise bout during each treatment session. Two-way ANOVAs will be used to examine the main effects of treatment and treatment-order interaction on pulse wave velocity, muscle cross-sectional area, perceptual responses, and exercise performance.

ELIGIBILITY:
Inclusion Criteria:

* Physically active (> 1,000 MET/min/wk) for at least six months. Weight stable for previous 6 months (+/-2.5 kg) Female subjects only- reported regular menstrual cycles for the last 2 years

Exclusion Criteria:

1. BP>140/90 mmHg
2. BMI>40 kg/m2
3. Diabetes
4. Familial hypercholesterolemia
5. Past or current history of CHD, stroke or major CVD events. Respiratory diseases (not including asthma), endocrine or metabolic, neurological, or hematological disorders that would compromise the study or the health of the subject.
6. Women must not be pregnant, plan to become pregnant during the study, or be nursing
7. Active renal or liver disease
8. All medications and supplements that influence dependent variables*
9. Recent surgery < 2 months
10. Alcohol abuse
11. Sleep apnea
12. Claustrophobia

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 27 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Arterial Stiffness | From enrollment to the end of treatment at 4 weeks
  Non-invasive pulse tonometers (Complior Analytic Tonometer, Alam Medical, Vincennes, France) will be used to simultaneously obtain arterial pressure waveforms at the carotid, brachial, radial and femoral arteries throughout ten cardiac cycles. Surface distance between the two recording sites will be measured to the nearest 0.5 cm. Subsequently, this process is repeated to measure arterial pressure waveforms at the carotid and radial arteries. Pulse wave velocity for the carotid-femoral (aortic PWV) and carotid-radial (brachial PWV) recordings will be determined by normalizing the waveform foot-to-foot time delay to the distance between recording sites (i.e., PWV = D (cm)/Δt (sec)). The participant will remain supine exactly as they were positioned during the tonometry acquisition sequence. An enlarged caliper will be used to measure the distance between the carotid and radial tonometer, and the distance between the carotid and femoral tonometer.

SECONDARY OUTCOMES:
Muscle Morphology | From enrollment to the end of treatment at 4 weeks
  Participants' muscle cross-sectional area (mCSA) and echo intensity (EI) of the vastus lateralis (VL) muscle will be assessed using a brightness mode (B-mode) of the ultrasound imaging system (Terason t3300, MA, USA) and a multi-frequency linear-array probe (Model 15L4 Smart Mark 4-15 MHz, 50-mm field of view). All ultrasonic scans will be conducted on the participants' right arm to measure the mCSA and EI of the VL. Each participant will be instructed to lay in a supine position with their shoulder abducted at 90 degree and elbow flexed at 90 degrees. The VL measurements will be obtained from their right leg at 50% of the distance between the greater tubercle and lateral epicondyle. Locations of measurements will be marked with indelible ink to ensure scans will be taken at the same area for all scans. During every scan, water soluble gel will be applied on the skin and ultrasound probe to maximize acoustic coupling and reduce near-field artifacts.

CONTACTS AND LOCATIONS:
Locations (1):
- Salisbury University, Salisbury, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Dissemination of data will occur after publication upon request.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: January 2026 - December 2029